CLINICAL TRIAL: NCT04526314
Title: Treatment and Outcomes of Stage III Colon Cancer in Patients 80 Years of Age and Older
Status: Completed | Type: Observational
Sponsor: Registre des Tumeurs Digestives du Finistère (Other)
Responsible Party: Sponsor
Other Study IDs: 908270
Record Dates: First submitted 2020-08-15; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Colon Adenocarcinoma
Keywords: stage 3 colon cancer; elderly; survival; surgery; chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stage 3 with adjuvant chemotherapy
  Interventions: Other: observational
- Stage 3 without adjuvant chemotherapy
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — observational

SUMMARY:
The objective of this study was to assess survival trends in elderly patients with stage III colon cancer

DETAILED DESCRIPTION:
This retrospective population-based study included patients aged 80 years and older with stage III colon adenocarcinoma who underwent surgery between 2007 and 2014.

ELIGIBILITY:
Inclusion Criteria:

• Stage 3 colon adenocarcinoma

Exclusion Criteria:

* Rectal tumors
* Patients receiving neo-adjuvant chemotherapy or radiotherapy
* Tumours of the appendix
* Tumours with histology other than adenocarcinoma

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: clinical data
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2007-2014
  months

CONTACTS AND LOCATIONS:
Overall Officials: Michel Robaskiewicz, MD PhD, Study Chair — REGISTRE DES TUMEURS DIGESTIVES DU FINISTERE
Locations (1):
- Registre de tumeurs digestives du Finistère, Brest, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badic B, Oguer M, Cariou M, Kermarrec T, Bouzeloc S, Nousbaum JB, Robaszkiewicz M, Queneherve L. Prognostic factors for stage III colon cancer in patients 80 years of age and older. Int J Colorectal Dis. 2021 Apr;36(4):811-819. doi: 10.1007/s00384-021-03861-6. Epub 2021 Feb 2. PMID 33528749